CLINICAL TRIAL: NCT00343369
Title: Multicentric Study for the Treatment of Children With Acute Lymphoblastic Leukemia
Brief Title: Combination Chemotherapy in Treating Young Patients With Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000455738; GER-COALL-07-03; EU-205104
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2006-06

CONDITIONS: Leukemia
Keywords: B-cell childhood acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Mercaptopurine; Methotrexate; pegaspargase; Prednisolone; Teniposide; Thioguanine; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: mercaptopurine
Drug: methotrexate
Drug: pegaspargase
Drug: prednisolone
Drug: teniposide
Drug: thioguanine
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating acute lymphoblastic leukemia.

PURPOSE: This randomized phase III trial is studying different combination chemotherapy regimens to compare how well they work in treating young patients with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose of daunorubicin hydrochloride that is equivalent to 30 mg/m² of doxorubicin hydrochloride in pediatric patients with acute lymphoblastic leukemia (ALL).
* Determine whether it is possible to reduce therapy in pediatric patients with low-risk ALL and a PVA (prednisolone-vincristine-asparaginase) score of 3+4 without loss of efficacy.
* Investigate the role of single nucleotide polymorphisms of infection defense gene for infectious complications during therapy in these patients.
* Reduce neurological complications by reducing doses of intrathecal methotrexate.
* Reduce allergic reactions against asparaginase (ASP) by using pegaspargase after E. coli ASP.

OUTLINE: This is a randomized, multicenter study.

* Prephase: Patients are randomized to 1 of 3 treatment arms.

  * Arm I: Patients receive doxorubicin hydrochloride IV once.
  * Arm II: Patients receive daunorubicin hydrochloride IV once.
  * Arm III: Patients receive daunorubicin hydrochloride IV once at a higher dose than in arm II.
* Induction phase: All patients receive vincristine IV 4 times weekly, daunorubicin hydrochloride IV 3 times weekly, and oral prednisolone daily for 4 weeks.
* Intensive phase: Patients are stratified according to risk (low vs high).

  * Low-risk disease*: Patients receive 4 courses of methotrexate IV and asparaginase intramuscularly (IM).
  * High-risk disease*: Patients receive 6 courses of cyclophosphamide IV, methotrexate IV, and asparaginase IM.

All patients also receive methotrexate IV, teniposide IV, cytarabine IV, high-dose cytarabine IV, and asparaginase IM after completion of the above regimen.

* CNS phase: All patients receive intrathecal (IT) methotrexate for 3 doses and oral mercaptopurine for 4 weeks. Patients with T-cell acute lymphoblastic leukemia or patients who have blasts in cerebrospinal fluid at diagnosis or whose WBC > 200/nL at diagnosis OR whose WBC between 100-200/nL at diagnosis and blasts > 1/nL after prephase chemotherapy undergo cranial irradiation.
* Reinduction phase: Patients are stratified according to risk (low vs high)

  * Low-risk disease*: Patients receive 2 courses of doxorubicin hydrochloride IV, vincristine IV, and oral dexamethasone; pegaspargase IM once; and 1 course of cyclophosphamide IV, cytarabine IV, and oral thioguanine.
  * High-risk disease*: Patients receive 4 courses of doxorubicin hydrochloride IV, vincristine IV, and oral dexamethasone; pegaspargase IM twice; and 2 courses of cyclophosphamide IV, cytarabine IV, and oral thioguanine.
* Maintenance phase: All patients receive oral mercaptopurine daily and methotrexate IV once weekly for up to 2 years after diagnosis.

NOTE: *In addition to those defined in Disease Characteristics, patients who do not achieve remission after induction phase are treated as high-risk disease, patients who achieve remission after induction phase are treated as low-risk disease

PROJECTED ACCRUAL: A total of 550 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with acute B-precursor or T-cell acute lymphoblastic leukemia (ALL)
* Meets 1 of the following risk criteria:

  * Low-risk disease, defined by any of the following:

    * WBC < 25/nL
    * B-precursor ALL

      * Excluding pro-B ALL
  * High-risk disease, defined by any of the following:

    * WBC ≥ 25/nL
    * T-cell ALL or pro-B ALL
    * Chromosomal translocation 4/11

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* More than 7 days since prior therapy with steroids, vincristine, or daunorubicin hydrochloride
* More than 7 days since prior cytotoxic therapy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 550 (Estimated)
Dates: Start 2003-01

PRIMARY OUTCOMES:
Dose of daunorubicin hydrochloride that is equivalent to 30 mg/m² of doxorubicin hydrochloride
Reduce therapy in low-risk patients without loss of efficacy
Reduce neurological complications
Reduce allergic reactions against asparaginase

CONTACTS AND LOCATIONS:
Overall Officials: Gritta Janka-Schaub, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (16):
- Germany (16):
  - Evangelisches Krankenhauus Bielfeld, Biefeld
  - Klinikum Bremen-Mitte, Bremen
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitats - Kinderklinik, Greiswald
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Kreskrankenhaus Kinderabteilung, Heide
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Klinikum Krefeld GmbH, Krefeld
  - Universitaets - Kinderklinik, Leipzig
  - Johannes Gutenberg University, Mainz
  - Krankenhaus Neuwerk Klinik fuer Kinder und Jugendmedizin, Mönchengladbach
  - Dr. von Haunersches Kinderspital der Universitaet Muenchen, Munich
  - Staedtisches Krankenhaus Muenchen - Harlaching, Munich
  - Klinik St. Hedwig-Kinderklinik, Regensburg
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Helios Kliniken Wuppertal University Hospital, Wuppertal